CLINICAL TRIAL: NCT05929846
Title: Back to Living Well: Implementation of a Community-based Program for the Secondary and Tertiary Prevention of Low Back Pain
Brief Title: Back to Living Well: Implementation of a Community-based Program for Low Back Pain
Status: Active, not recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Luciana Macedo, Principal Investigator, McMaster University
Other Study IDs: 15354
Record Dates: First submitted 2023-06-05; First posted 2023-07-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In-Person: Participants will be assessed by a LiveWell specialist to assess functional goals and baseline capacity and design an individualized program. LiveWell specialist may also refer participants for an assessment with a physiotherapist based on a pre-defined criteria including redflag for serious conditions. Participants will engage in a 12-week program consisting of 45 minute sessions 3 times a week. Day 1 will include individualized program at the fitness center, Day 2 will include a group class exercises ending with mindfulness activities, action planning and education. Day 3 will consist of an independent day when participants can attend other classes at the YMCA or repeat the fitness center. In addition, there will be 12 virtual videos of education on self-management that will be discussed during the group activity day (Day 2) .
  Interventions: Other: Back to Living Well Program
- e-Health: Participants will be assessed by a LiveWell specialist to assess functional goals and baseline capacity and provide recommendation on exercise modifications and the program. LiveWell specialist may also refer participants for an assessment with a physiotherapist based on a pre-defined criteria including redflag for serious conditions. Participants will engage in a 12-week program consisting of 45 minute sessions 3 times a week. They will be provided with 3 exercise videos (including 3 levels of exercises per video) and will also have access to the on-demand YMCA platform for additional videos. In addition, there will be 12 virtual videos of education on self-management that will be discussed during follow-up phone calls. Participants will also be provided with an action planning document to complete at home. All online participants will have a phone call with the LiveWell specialist at 3 and 7 weeks to discuss the program, action planning and the education materials.
  Interventions: Other: Back to Living Well Program

INTERVENTIONS:
Other: Back to Living Well Program — The Back to Living Well program (BLW), a sustainable community-based program for persons with persistent mild to moderate LBP. The goal of the intervention is to provide an opportunity for community dwelling persons with persistent mild to moderate LBP to learn how to safely engage in exercise and become active self-managers. The 12-week program will engage participants in weekly exercise sessions, education and self management sessions, and encourage independent exercise at least 1x per week. All participants will be encouraged to complete an action plan and watch online education videos weekly.

SUMMARY:
Low back pain (LBP) is usually a long-term condition with episodes of improvement, remission, and recurrence. There is evidence that long term exercise combined with education and self-management is effective at reducing the negative consequences of LBP. However, problems with uptake and long-term adherence to such programs are often reported in the literature. Using best available evidence, the implementation of the BackToLivingWell (BLW) will be evaluated, a community-based online or in-person program for the prevention long term disability due to LBP through exercise and self management.

DETAILED DESCRIPTION:
The study will evaluate the implementation of The Back to Living Well program (BLW), a sustainable community-based program for persons with persistent mild to moderate LBP. The goal of the intervention is to provide an opportunity for community dwelling persons with persistent mild to moderate LBP to learn how to safely engage in exercise and become active self-managers. Through the engagement in exercise and healthy lifestyle behaviours, the program aims to prevent activity-limiting flares as well as minimize the ongoing impact of the condition with improvements in function and quality of life.

Persons with LBP will be invited to participate in either the in-person or e-health program based on their choices. We will conduct a mixed-method study with a quantitative and a qualitative portion. This will include participants completing the program and questionnaires at baseline, 3-, 6- and 12- months, as well as longitudinal qualitative interviews at the same time points to assess: 1) barriers and facilitators to the program, 2) factors that contribute to negative and positive responses to the program. This may include how intervention outcomes are related to the program, personal and societal factors, and 3) factors that influence the selection of in-person versus online intervention.

In addition, to evaluate symptom trajectories, an ecological Momentary Assessment (EMA) will be collecting data over the same time points (baseline, 3-, 6- and 12- months). Weekly outcomes will be collected for 1-year using a smartphone application. The results of this study will provide evidence to inform future implementation of the program including strategies that could lead to better outcomes. Additionally, LiveWell specialists delivering the program and YMCA staff will be interviewed at the end of the program.

Overall, the RE-AIM framework will be used to guide our implementation. Additionally, using the Theoretical Domains Framework, the Technology Acceptance Model and the Neuromatrix Model of Pain we will construct a theory-based approach to:

1. Identify program barriers and facilitators from the perspective of the patients,
2. Identify factors contributing to negative and positive outcomes as well as outcome trajectories, including how outcomes are related to the program, personal and contextual factors and,
3. Identify factors influencing participants to select an in-person or e-health program,
4. Evaluation program specific implementation barriers and facilitators from the perspectives of the organization and care delivery perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Currently starting or enrolled in the Back to Living Well program at a YMCA in Downtown Hamilton, Les Chater, Ron Edwards, Laurier Brantford or Flamborough
* Have non-specific LBP
* History of persistent LBP for 3 or more months that is mild, moderate, or severe
* If moderate levels of pain or less (pain <6) they must have a history of flares or at least one flare within the previous year, if pain >=6, flare is not necessary.
* 18 years old or older

Exclusion Criteria:

* Co-morbidity preventing participation in exercise based on screening using the Physical Activity Readiness Questionnaire and later not cleared by their family physician
* Inadequate English to complete questionnaires and interviews
* Participants who are currently seeking care for LBP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be individuals from the community suffering from LBP. We will recruit participants that have demonstrated interested on the Back to Living Well program and have reached out to the YMCA to learn more about the program and to register. Participants will be referred to the study by the YMCA at the time that they decide to enroll in the program in one of the YMCA available locations ( YMCA location in Downtown Hamilton, Les Chater, Ron Edwards, Laurier Brantford or Flamborough ) .
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | 12-months
  RMDQ is for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. The score ranges from 0 (no disability) to 24 (maximum disability).

SECONDARY OUTCOMES:
Pain NRS | Baseline, 3 months, 6 months & 12 months
  Average pain over the last week on a scale of 0 (no pain) to 10 (extreme pain).
Self Report Flare | Once a week for 12 months (week 0-week 52)
  Participants will meet the criteria for activity-limiting flare if pain has increased at least 2 points on a NRS- 10 point scale (MCID) over the previous week
Activity Limitation | Once a week for 12 months (week 0-week 52)
  Scale from 1-5 about the level in which pain interfered with day to day activities
EQ-5D-5L | Once a week for 12 months (week 0-week 52)
  Anxiety and Depression dimensions only. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  Depending on the level, a number is assigned to each dimension, so that a 5-digit number combination is obtained into a EQ5D Health State.
TAMPA Scale of Kinesiophobia | Baseline, 3 months, 6 months & 12 months
  a 17 item scale originally developed to measure the fear of movement related to chronic lower back pain.
Pain Self-Efficacy Questionnaire | Baseline, 3 months, 6 months & 12 months
  10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain.
Coping Strategies Questionnaire | Baseline, 3 months, 6 months & 12 months
  5 item scale to measure ability to cope with pain. Minimum score of 0 and maximum score of 36, with higher scores indicating greater use of a particular coping strategy.
Pain Catastrophizing Scale | Baseline, 3 months, 6 months & 12 months
  13-item self report measure designed to assess catastrophic thinking related to pain A total score ranges from 0-52, with higher scales representing higher pain catastrophizing for individuals with chronic pain.
EQ-5D-5L | Baseline, 3 months, 6 months & 12 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  Depending on the level, a number is assigned to each dimension, so that a 5-digit number combination is obtained into a EQ5D Health State.
  The EQ VAS score is rated on a scale of 0-100 points. 0 points correspond to the worst possible health status, while 100 points correspond to the best possible health status.
International Physical Activity Questionnaires | Baseline, 3 months, 6 months & 12 months
  27-item self-reported measure of physical activity for use with individual adult patients. There are two forms of output from scoring the IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Patient Specific Functional Scale | Baseline, 3 months, 6 months & 12 months
  The PSFS is a self-reported valid, reliable, and responsive outcome measure for patients with back, neck, knee and upper extremity problems. Participants identify 3 important activities that you are unable to do or have difficulty performing. Patients are asked to rate (on an 11-point scale) the current level of difficulty associated with each activity. 0" represents "unable to perform" and "10" represents "able to perform at prior level"
PROMIS IMPACT | Baseline, 3 months, 6 months & 12 months
  An adapted version of this survey will collect data on back pain.
Treatment Self Regulation Questionnaire | Baseline, 3 months, 6 months & 12 months
  This self-reported questionnaire assesses the degree to which a person's motivation for the health behaviors. Likert typescale ranging from 1 (not at all true) to 7 (very true). There are three subscales to the scale: the autonomous regulatory style; the controlled regulatory style; and amotivation (which refers to being unmotivated).
Center for Epidemiologic Studies Depression Scale | Baseline, 3 months, 6 months & 12 months
  A 20-item measure self reported scale to measure depressive symptoms. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Exercise Adherence Rating Scale | Baseline, 3 months, 6 months & 12 months
  A 6-item questionnaire aimed at measuring adherence behavior and exploring reasons for nonadherence. The six items are scored using an ordinal answer scale (0 = strongly agree to 4 = totally disagree), with higher scores indicating greater adherence (0 to 24).
Adherence exercise | After completion of the program (3 months)
  Number of exercise session attended or exercise videos watched as per online program
Adherence education | After completion of the program (3 months)
  Number of virtual education videos watched

OTHER OUTCOMES:
Long term physical activity | 12 months after baseline
  Length of YMCA membership

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Macedo, PhD, Principal Investigator — McMaster University; Julie Richardson, PhD, Principal Investigator — McMaster University; Joy MacDermid, PhD, Principal Investigator — McMaster University; Mark Hancock, PhD, Principal Investigator — Macquarie University; Michele Crites Battie, Principal Investigator — Western University; Bruno Saragiotto, PhD, Principal Investigator — Universidade Cidade de Sao Paulo; Jill Hayden, PhD, Principal Investigator — Dalhousie University; Alison Rushton, EdD, Principal Investigator — Western University; Tara Packham, PhD, Principal Investigator — McMaster University; Steven Bray, PhD, Principal Investigator — McMaster University; Meridith Griffin, PhD, Principal Investigator — McMaster University; Diego Silva, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Macedo L, Di Pelino S, Santos VS, Richardson J, MacDermid J, Hancock M, Battie MC, Saragiotto BT, Hayden JA, Rushton A, Packham T, Freman M, Bray S, Griffin M, Hladysh G, Miller P, Attwell S. Implementation of back to living well, a community-based program for the tertiary prevention of low back pain: a study protocol. BMC Musculoskelet Disord. 2024 Jul 27;25(1):593. doi: 10.1186/s12891-024-07712-7. PMID 39068385